CLINICAL TRIAL: NCT03834389
Title: The Effect of Case-Based Learning Method on Perceived Competence and Critical Thinking Levels in Nursing Students: Mixed Method
Brief Title: The Effect of Case-Based Learning Method on Perceived Competence and Critical Thinking Levels
Acronym: Case-Based
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Rukiye Burucu, Doctorate student, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RBurucu
Record Dates: First submitted 2018-08-30; First posted 2019-02-08 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-01

CONDITIONS: Educational Problems
Keywords: case- based learning; critical thinking; self-efficacy; nursing education; nursing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Experimental group: case-based teaching method applied
  Interventions: Behavioral: Case- based Learning
- Control Group (No Intervention): Control group: classical teaching method applied

INTERVENTIONS:
Behavioral: Case- based Learning — critical thinking, self efficacy, focus group interview
  Arms: Experimental Group

SUMMARY:
Second-year nursing students are randomly assigned to experimental and control groups. The case-based teaching method was applied to the experimental group and the classical teaching method was applied to the control group. After the initiative, both groups observed differences in perceived competence and critical thinking levels. In addition, the focus groups were interviewed with the experimental group and the opinions and suggestions about the initiative were evaluated qualitatively and the total mix method was used.

DETAILED DESCRIPTION:
Nursing secondary school students were randomized into two groups. Case-based training was given to the experimental group, and classical training was given to the control group. Critical thinking scale and self-efficacy scale both before and after the training were applied to both groups. Posttest scores were calculated and compared for both groups. The focus group consultation with 10 people from the experimental group was carried out and the opinions and suggestions about the initiative were taken and evaluated. Permission was obtained in writing from all institutions before and after the participants, and the study was conducted by creating ethical conditions.Four separate training cases were given to the experimental group. the control group continued the classical training and no intervention was made.

ELIGIBILITY:
Inclusion Criteria:

* Become a nursing 2nd year student
* Want to participate in the research
* Not to be in the health profession
* Having passed the course of internal medicine nursing
* Being the first to see the surgical diseases nursing course
* Be able to devote time for case discussions outside of class

Exclusion Criteria:

- Being a foreign national (Unable to speak / understand Turkish effectively)

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
CRITICAL THINKING TENDENCY SCALE | 4 months
  It was developed by a Turkish researcher and reliability of validity was done. The scale covers 49.161% of the variance. Factor loads range from 0.33 to 0.71. Sub-dimensions: metacity, flexibility, systematicness, determination and patience, open mindedness. The scale consists of 49 questions in total. Scale your scale; I totally agree (5), I mostly agree (4), Partially agree (3), I mostly do not agree (2), I never agree (1). The test retest correlation coefficient of the scale was 0.761 and the correlation coefficient between the two half scores was 0.95. The Cronbach Alpha coefficient is 0.963. Confirmatory factor analysis was performed with the AMOS program (Ratio = 2778.981, Sd = 1073, X2 / Sd = 2.590, GFI = 0.903, CFI = 0.932, RMSEA = 0.038). The total score ranges from 49 to 245, with a high score indicating a high tendency to think critically
Effect of case-based learning method on self-efficacy level | 4 months
  The German version was originally used by Schwarzer. It was originally prepared as 20 items, then reduced to 10 items. Over time, it has been translated and used in more than twenty languages. Item total correlations are between 0.30 and 0.77. Reliability of Turkish validity was done; Alpha internal consistency coefficient was 0.79-0.63, total alpha coefficient was 0.83. Test-retest reliability coefficient of the scale is r = 0.80, p <0.001. Factor analys's results of the Turkish version show that it accounts for 47% of the total variance. The item total score correlation coefficients are between 0.37 and 0.59. The items of the scale have scores ranging from 1 to 4, with a total score ranging from 10 to 40. High score is considered as high self-efficacy perception.

SECONDARY OUTCOMES:
Focus group interview | 4 months
  Group suggestions and comments (qualitative study)

CONTACTS AND LOCATIONS:
Locations (1):
- Selçuk Univercity, Konya, Selçuklu/Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
it is planned that the work will be shared after the writing is completed